CLINICAL TRIAL: NCT03912545
Title: Evaluation of the Clinical Performance of the Quantra System With the QStat Cartridge in Trauma and Obstetric Hemorrhage
Brief Title: Evaluation of the Clinical Performance of the Quantra System With the QStat Cartridge
Status: Completed | Type: Observational
Sponsor: HemoSonics LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: HEMCS-019
Record Dates: First submitted 2019-04-09; First posted 2019-04-11 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Blood Loss Massive; Trauma; Hemorrhage, Postpartum
Keywords: Viscoelastic testing; Coagulation; Quantra; Hemostasis
MeSH Terms: conditions — Wounds and Injuries; Postpartum Hemorrhage; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Trauma patients: Subjects experiencing major trauma such that viscoelastic testing is performed as standard of care to assess coagulopathy.
  Interventions: Diagnostic Test: Quantra System
- Obstetric hemorrhage patients: Subjects experiencing obstetric hemorrhage such that viscoelastic testing is performed as standard of care is performed to assess coagulopathy.
  Interventions: Diagnostic Test: Quantra System

INTERVENTIONS:
Diagnostic Test: Quantra System — Diagnostic device to monitor coagulation properties of a whole blood sample at the point-of-care.
  Other Names: Quantra QStat Cartridge

SUMMARY:
This pilot study will evaluate the performance of the Quantra System comprised of the Quantra Hemostasis Analyzer with the QStat Cartridge in trauma patients or patients with OB hemorrhage.

DETAILED DESCRIPTION:
The Quantra System is a fully integrated and automated in vitro diagnostic device which uses SEER Sonorheometry, an ultrasound-based technology, to characterize the viscoelastic properties of a whole blood sample during coagulation. The QStat Cartridge was developed to monitor hemostasis in patients that may experience a range of coagulopathies of various etiologies including fibrinolytic defects. These patients include the trauma and obstetric hemorrhage populations. The cartridge consists of four independent channels each containing different sets of reagents, which provide four measurements performed in parallel yielding five parameters that depict the functional status of a patient's coagulation system.

This single-center, prospective, observational pilot study will evaluate the performance of the Quantra System with the QStat Cartridge as compared to standard coagulation tests and comparable measures using conventional viscoelastic testing methods.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥ 18 years of age
* Subject has one of the following conditions and is a candidate for a ROTEM test to be performed to access coagulopathy: trauma patient; patient with OB hemorrhage.

  * For trauma patients; subject must be experiencing major trauma (preferably requiring the highest level of team activation) with active bleeding or deemed at high risk of significant bleeding according to mechanism of injury.
  * For subjects experiencing OB hemorrhage, one of the following conditions must be met (to be confirmed):

    * Estimated blood loss during vaginal delivery is greater than 1000 mL
    * Estimated blood loss during cesarean delivery is greater than 1500 mL
    * Placental abruption with hemorrhage of any quantity blood loss
    * Clinically suspected disseminated intravascular coagulation (DIC)
    * Is under consideration for administration of tranexamic acid (TXA) for treatment of hemorrhage.
* Subject is willing to participate, and is willing to consent (either prospectively or by deferred consent)

Exclusion Criteria:

* Subject is younger than 18 years of age
* Subject is known to have received antifibrinolytic therapy immediately prior to presentation to trauma unit or during labor just prior to OB hemorrhage.
* Subject is unable to provide written informed consent (either prior to performing any study related procedures or by deferred consent)
* Subject is currently enrolled in a distinct study that might confound the results of the proposed study
* Subject is affected by a condition that, in the opinion of the clinical team, may pose additional risks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential study participants will be adult (>18 years) trauma patients or patients with OB hemorrhage such that viscoelastic testing is performed as standard of care to assess coagulopathy.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2019-07-11 (Actual); Study Completion 2019-07-11 (Actual)

PRIMARY OUTCOMES:
Comparison of Quantra Clot Time and Clot Stiffness results to standard coagulation test results | Upon arrival to emergency department (trauma subjects) or upon presentation with obstetric hemorrhage, prior to the administration of blood products or antifibrinolytics in parallel with samples collected for routine ROTEM analysis and laboratory assays
  Coagulation function assessed by Quantra and standard coagulation tests
Comparison of Quantra Clot Time and Clot Stiffness results to ROTEM Delta results | Upon arrival to emergency department (trauma subjects) or upon presentation with OB hemorrhage, prior to the administration of blood products or antifibrinolytics in parallel with samples collected for routine ROTEM analysis and laboratory assays
  Coagulation function assessed by Quantra and ROTEM Delta
Comparison of Quantra Fibrinolysis results to ROTEM Delta results | Upon arrival to emergency department (trauma subjects) or upon presentation with OB hemorrhage, prior to the administration of blood products or antifibrinolytics in parallel with samples collected for routine ROTEM analysis and laboratory assays
  Coagulation function assessed by Quantra and ROTEM Delta

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Tech University Health Sciences Center El Paso, El Paso, Texas, United States

IPD SHARING:
Plan to Share IPD: No